CLINICAL TRIAL: NCT00887614
Title: Mechanisms of Mindfulness: Effects on Sleep Quality, Stress Physiology and CVD Risk
Brief Title: Mindfulness, Emotional Well-being, and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jeffrey M. Greeson, PhD, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002861; 5K99AT004945-02 (NIH)
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Stress, Psychological; Sleep
Keywords: mindfulness; meditation; stress; rumination; emotion regulation; sleep quality; spirituality; quality of life
MeSH Terms: conditions — Stress, Psychological; Rumination Syndrome; Emotional Regulation; Sleep Initiation and Maintenance Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MBSR (Experimental): Participation will involve online completion of a questionnaire survey before and after the Mindfulness-Based Stress Reduction (MBSR) intervention. Specifically, research study participants will complete validated self-report measures to assess mindfulness, cognitive-emotional processes, sleep quality, symptoms of stress, sense of spirituality, and quality of life before and after the MBSR intervention.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — The MBSR program consists of 8 weekly classes that last for 2.5 hours each and a commitment to daily meditation practice for the duration of the course. Classes include didactic instruction on mindfulness and its relationship to stress and health, guided meditation practices, and group discussion. Mindfulness meditation practices include awareness of breathing, awareness of emotions, body scan, mindful hatha yoga, mindful walking, mindful eating, mindful listening, and lovingkindness (metta). Participants are expected to practice formal meditation outside of class for 20-45 min per day, 6 days per week. In addition, participants are encouraged apply mindfulness to everyday activities like eating, communicating with others, and hobbies. Written materials and audio CDs with guided meditations and yoga are provided. The course also includes one full day (7-hours) of meditation on a Saturday following the 6th week of class.

SUMMARY:
The purpose of this study is to determine whether participating in a Mindfulness-Based Stress Reduction (MBSR) program increases mindful attention and awareness, and whether anticipated changes in mindfulness relate to improved emotional well-being, sleep quality, physical symptoms of stress, sense of spirituality, and quality of life following MBSR.

DETAILED DESCRIPTION:
This study will be conducted among men and women participating in 8-week Mindfulness-Based Stress Reduction (MBSR) classes at Duke Integrative Medicine in Durham, North Carolina. The central hypothesis of this NIH-funded clinical trial (K99 AT004945, PI: Greeson) is that mindfulness meditation training is associated with increased levels of mindfulness and improved cognitive-emotional functioning that, together, are associated with reduced psychological distress, improved sleep quality, and decreased stress-related physical symptoms, including muscle tension, headache, and gastrointestinal complaints. This study is designed to examine psychological mechanisms that may explain individual differences in MBSR outcomes. This knowledge is important because it will help us better understand who is most likely to benefit from mindfulness meditation training, and why. The results from this study are expected to elucidate mechanisms underlying the mental and physical health benefits of stress reduction, which can help guide clinicians in referring the most suitable patients to local MBSR programs.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in a self-pay MBSR course at Duke Integrative Medicine
* Must be able to speak and read English

Exclusion Criteria (Apply to Duke's MBSR program, and thus to the research study):

* Active substance abuse/dependence
* Severe mental illness
* Difficulty being redirected to task in a group setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Mindfulness | 2 months
  Attention to and awareness of thoughts and feelings.

SECONDARY OUTCOMES:
Sleep quality | 2 months
  Self-reported sleep quality during the past month, as indicated by sleep latency (time to fall asleep), subjective sleep quality (very good, fairly good, fairly bad, very bad), sleep duration (hours of sleep per night), sleep efficiency (# of hrs asleep/# of hrs in bed), use of sleep medication, and daytime functioning (mental clarity and energy/fatigue).
Cognitive perseveration | 2 months
  Forms of distressing repetitive thought, including unwanted intrusive thoughts and rumination.
Emotion regulation | 2 months
  Strategies to regulate emotions, including suppression, reappraisal, and avoidance.
Spirituality | 2-months
  Ordinary experiences of connection with the transcendent in daily life.
Health-related quality of life | 2-months
  Mental and physical functioning and well-being during daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Greeson, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Integrative Medicine, Durham, North Carolina, United States

REFERENCES:
- [Background] Greeson JM. Mindfulness Research Update: 2008. Complement Health Pract Rev. 2009 Jan 1;14(1):10-18. doi: 10.1177/1533210108329862. PMID 20047019
- [Result] Greeson JM, Webber DM, Smoski MJ, Brantley JG, Ekblad AG, Suarez EC, Wolever RQ. Changes in spirituality partly explain health-related quality of life outcomes after Mindfulness-Based Stress Reduction. J Behav Med. 2011 Dec;34(6):508-18. doi: 10.1007/s10865-011-9332-x. Epub 2011 Mar 1. PMID 21360283
- See also: Website for the Mindfulness-Based Stress Reduction (MBSR) program at Duke Integrative Medicine — http://www.dukeintegrativemedicine.org/index.php/2009012037/classes-workshops-events/mindfulness-based-stress-reduction.html
- See also: Free full-text version of "Mindfulness Research Update:2008" — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2679512/pdf/nihms107164.pdf